CLINICAL TRIAL: NCT00401726
Title: Patient Outcomes With Education, Drug Therapy, and Support (POETS): A Multicenter, Open-label, Randomized Study to Evaluate Depressed Subjects Treated With Venlafaxine Extended-release vs. Venlafaxine Extended-release Plus the Dialogues Time to Talk Program in a Primary Care Setting
Brief Title: Open-Label, Randomized Study Evaluating Treatment With Venlafaxine Extended-Release Plus Dialogues Time to Talk Program
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0600B1-416
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Results first posted 2010-06-29 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Depressive Disorder, Major
Keywords: Major Depressive Disorder; Depression; Anxiety
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Anxiety Disorders

INTERVENTIONS:
Drug: Venlafaxine ER
Behavioral: Dialogues Time to Talk Program

SUMMARY:
The purpose of this study is to evaluate the effect of the Dialogues Time to Talk program in subjects treated with Venlafaxine Extended Release (ER). Dialogues Time to Talk Program is a patient management program, which aims to help patients achieve successful outcomes by reinforcing physician treatment efforts, providing feedback to treating physicians, and encouraging better physician-patient communications.

ELIGIBILITY:
Inclusion Criteria:

* Currently experiencing a major depressive episode, which requires the initiation of antidepressant drug treatment or a change in current antidepressant drug treatment
* At least 18 years of age

Exclusion Criteria:

* History or presence of bipolar disorder
* Current treatment with venlafaxine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 537 (Actual)
Dates: Start 2006-06; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (42):
- United States (42):
  - Birmingham, Alabama
  - Mesa, Arizona
  - Little Rock, Arkansas
  - San Jose, California
  - Avon, Connecticut
  - Cromwell, Connecticut
  - Wilmington, Delaware
  - Ocala, Florida
  - Pinellas Park, Florida
  - Stuart, Florida
  - Atlanta, Georgia
  - Cartersville, Georgia
  - Rome, Georgia
  - Idaho Falls, Idaho
  - Newburgh, Indiana
  - Waterloo, Iowa
  - Metairie, Louisiana
  - Benzonia, Michigan
  - Interlochen, Michigan
  - Kalamazoo, Michigan
  - Chesterfield, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Kettering, Ohio
  - Mason, Ohio
  - Mogadore, Ohio
  - Allentown, Pennsylvania
  - Newtown, Pennsylvania
  - Reading, Pennsylvania
  - Warwick, Rhode Island
  - Anderson, South Carolina
  - Greer, South Carolina
  - Bristol, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Charleston, West Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in the United States from June 2006 to March 2007.
Pre-assignment Details: Subjects were enrolled according to the inclusion / exclusion criteria. There was not a screening period.
Groups:
- Venlafaxine Extended Release (ER): 75-225 mg per day
- Venlafaxine Extended Release (ER) Plus Dialogues: Venlafaxine ER 75-225 mg per day plus "Dialogues Time to Talk" program (Dialogues). Dialogues is a patient management program designed to reinforce physician treatment efforts, provide feedback to treating physicians and encourage better physician-patient communication.
Period: Overall Study
Arm/Group | Venlafaxine Extended Release (ER) | Venlafaxine Extended Release (ER) Plus Dialogues
Started | 269 | 268
Completed | 172 | 156
Not Completed | 97 | 112
Not completed — Adverse Event | 34 | 45
Not completed — Death | 0 | 3
Not completed — Sponsor Request | 0 | 1
Not completed — Physician Decision | 3 | 6
Not completed — Lost to Follow-up | 23 | 20
Not completed — Protocol Violation | 6 | 3
Not completed — Withdrawal by Subject | 18 | 24
Not completed — Lack of Efficacy | 4 | 6
Not completed — Protocol Deviation | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Venlafaxine Extended Release (ER) | Venlafaxine Extended Release (ER) Plus Dialogues | Total
Number analyzed (Participants) | 269 | 268 | 537
Age Continuous [Mean (Standard Deviation); unit: years] | 44.13 (13.59) | 45.25 (13.83) | 44.69 (13.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199 | 190 | 389
  Male | 70 | 78 | 148

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Responding "Very Satisfied" on Satisfaction With Depression Care Scale (SDCS)
Description: Patient satisfaction with depression care treatment was evaluated by patient self-assessment using the SDCS, a 10-point visual analog scale (0=not at all satisfied, 10=extremely satisfied). "Very satisfied" was defined as a score of greater than or equal to 8.
Time Frame: 112 days
Population: The analysis population was the Modified Intent to Treat population, which included all patients who received a prescription and had at least 1 post-baseline efficacy evaluation; last observation carried forward.
Measure: Number; unit: participants
Arm/Group | Venlafaxine Extended Release (ER) | Venlafaxine Extended Release (ER) Plus Dialogues
Number analyzed (Participants) | 254 | 239
participants | 160 | 138
Statistical Analysis 1: Comparison: Venlafaxine Extended Release (ER) vs Venlafaxine Extended Release (ER) Plus Dialogues; Test type: Superiority or Other; p = 0.218, Chi-squared; Risk Difference (RD) = 5.25

2. Secondary Outcome: Change in 17-item Hamilton Depression Scale Score From Baseline to 16 Weeks
Description: HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Items are scored on a 0 to 2 or 4 scale (0 = none/absent and 4 = most severe) with a maximum total score of 50. Change = 16 week adjusted mean HAM-D17 score minus baseline.
Time Frame: Baseline and 112 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Venlafaxine Extended Release (ER) | Venlafaxine Extended Release (ER) Plus Dialogues
Number analyzed (Participants) | 254 | 239
units on scale | -10.87 (0.39) | -11.03 (0.40)
Statistical Analysis 1: Comparison: Venlafaxine Extended Release (ER) vs Venlafaxine Extended Release (ER) Plus Dialogues; Test type: Superiority or Other; p = 0.76, ANCOVA; Mean Difference (Net) = 0.16, 95% CI [-0.92 to 1.25]

3. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) Score
Description: PGI-I is a global rating scale that measures disease improvement. Using a 7-point scale (1=very much improved, 7=very much worse), the patients rate how much their illness has improved or worsened relative to their baseline status.
Time Frame: 112 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Venlafaxine Extended Release (ER) | Venlafaxine Extended Release (ER) Plus Dialogues
Number analyzed (Participants) | 254 | 239
units on scale | 2.33 (0.08) | 2.51 (0.09)
Statistical Analysis 1: Comparison: Venlafaxine Extended Release (ER) vs Venlafaxine Extended Release (ER) Plus Dialogues; Test type: Superiority or Other; p = 0.148, ANCOVA; Mean Difference (Net) = -0.17, 95% CI [-0.41 to 0.06]

4. Secondary Outcome: Change in WHO 5-item Well Being Index Score From Baseline to 16 Weeks
Description: WHO 5-item Well Being Index (WHO-5) evaluates positive psychological well-being. WHO-5 consists of 5 questions and each is rated on a 6-point scale. The total score ranges from 0 to 25 (0=worst possible quality of life, 25=best possible quality of life). Change = 16 week adjusted mean WHO-5 score minus baseline.
Time Frame: Baseline and 112 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Venlafaxine Extended Release (ER) | Venlafaxine Extended Release (ER) Plus Dialogues
Number analyzed (Participants) | 254 | 239
units on scale | 6.86 (0.35) | 6.97 (0.36)
Statistical Analysis 1: Comparison: Venlafaxine Extended Release (ER) vs Venlafaxine Extended Release (ER) Plus Dialogues; Test type: Superiority or Other; p = 0.829, ANCOVA; Mean Difference (Net) = -0.11, 95% CI [-1.09 to 0.87]

5. Secondary Outcome: Number of Patients Compliant With Therapy
Description: Patient compliance with therapy was assessed using a Medical Adherence Questionnaire (MAQ). MAQ consisted of 5 levels of compliance with taking medicine: Never miss, Sometimes miss, Miss half of the time, Miss most of the time, Always miss. Compliance with therapy was defined as a response of "Never miss" or "Sometimes miss".
Time Frame: 112 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Venlafaxine Extended Release (ER) | Venlafaxine Extended Release (ER) Plus Dialogues
Number analyzed (Participants) | 254 | 239
participants | 248 | 232
Statistical Analysis 1: Comparison: Venlafaxine Extended Release (ER) vs Venlafaxine Extended Release (ER) Plus Dialogues; Test type: Superiority or Other; p = 0.728, Chi-squared; Risk Difference (RD) = 0.57

6. Secondary Outcome: Change in Inventory of Depressive Symptomatology - Self-Report (IDS-SR) Score From Baseline to 16 Weeks
Description: IDS-SR is a patient self-administered tool used to measure the severity of depressive symptoms. Each symptom is assessed on a scale of 0 to 3 (0=absence of symptom to 3=sever symptom) for a total maximum score of 84.
Time Frame: Baseline and 112 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Venlafaxine Extended Release (ER) | Venlafaxine Extended Release (ER) Plus Dialogues
Number analyzed (Participants) | 254 | 239
units on scale | -17.75 (0.71) | -17.50 (0.73)
Statistical Analysis 1: Comparison: Venlafaxine Extended Release (ER) vs Venlafaxine Extended Release (ER) Plus Dialogues; Test type: Superiority or Other; p = 0.805, ANCOVA; Mean Difference (Net) = -0.25, 95% CI [-2.24 to 1.74]

7. Secondary Outcome: Change in Sheehan Disability Scale Score From Baseline to 16 Weeks
Description: The Sheehan Disability Scale is a self-administered tool that measures functional impairment in 3 domains: Work/School, Social Life and Family Life/Home Responsibilities. The patient rates the extent to which each of these domains are impaired by his/her symptoms using a 10 point visual analog scale: (0=not at all impaired and 10=extremely impaired) for a total maximum score of 30.
Time Frame: Baseline and 112 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Venlafaxine Extended Release (ER) | Venlafaxine Extended Release (ER) Plus Dialogues
Number analyzed (Participants) | 254 | 239
units on scale | -7.99 (0.45) | -6.99 (0.47)
Statistical Analysis 1: Comparison: Venlafaxine Extended Release (ER) vs Venlafaxine Extended Release (ER) Plus Dialogues; Test type: Superiority or Other; p = 0.123, ANCOVA; Mean Difference (Net) = -1.0, 95% CI [-2.27 to 0.27]

8. Secondary Outcome: Number of Patients by Clinical Global Improvement - Global Improvement Score at 16 Weeks
Description: CGI-I is a global rating scale that measures disease improvement. Using a 7-point scale, the clinician rates how much the patient's illness has improved or worsened relative to the baseline status (1=very much improved, 7=very much worse).
Time Frame: 112 days
Population: The analysis population was the Modified Intent to Treat population, which included all patients who received a prescription and had at least 1 post-baseline efficacy evaluation; last observation carried forward. Data not available for one participant.
Measure: Number; unit: patients
Arm/Group | Venlafaxine Extended Release (ER) | Venlafaxine Extended Release (ER) Plus Dialogues
Number analyzed (Participants) | 253 | 239
patients
  CGI - 1 (very much improved) | 82 | 81
  CGI - 2 (much improved) | 84 | 75
  CGI - 3 (improved) | 50 | 49
  CGI - 4 (no change) | 24 | 21
  CGI - 5 (worse) | 11 | 8
  CGI - 6 (much worse) | 2 | 5
  CGI - 7 (very much worse) | 0 | 0
Statistical Analysis 1: Comparison: Venlafaxine Extended Release (ER) vs Venlafaxine Extended Release (ER) Plus Dialogues; CGI-I raw scores (range 1-7) analyzed by generalized Cochran-Mantel-Haenszel (CMH) test, stratified by study center using the ridit scoring option; Test type: Superiority or Other; p = 0.961, Cochran-Mantel-Haenszel; p-value based on comparison of mean score differences

ADVERSE EVENTS:
Arm/Group | Venlafaxine Extended Release (ER) | Venlafaxine Extended Release (ER) Plus Dialogues
Serious Adverse Events (participants affected / at risk) | 10/269 | 18/268
Other Adverse Events (participants affected / at risk) | 209/269 | 214/268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Venlafaxine Extended Release (ER) (N=269) | Venlafaxine Extended Release (ER) Plus Dialogues (N=268)
Accidental Injury (Injury, poisoning and procedural complications) | 1 | 1
Angina Pectoris (Cardiac disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular Accident (Vascular disorders) | 1 | 1
Chest pain (Cardiac disorders) | 0 | 1
Cholecystits (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Renal and urinary disorders) | 0 | 1
Coronary Artery Disorder (Cardiac disorders) | 0 | 2
Depression (Psychiatric disorders) | 1 | 0
Drug Abuse (General disorders) | 0 | 1
Hernia (General disorders) | 1 | 0
Hypertension (Cardiac disorders) | 0 | 1
Intracranial Hemorrhage (Vascular disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Neurosis (Psychiatric disorders) | 1 | 0
Non-specific Drug Reaction (General disorders) | 0 | 1
Overdose (General disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Self-injurious Ideation (General disorders) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 2
Suicide (Psychiatric disorders) | 0 | 1
Suicide Attempt (Psychiatric disorders) | 0 | 2
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
Thinking Abnormal (Psychiatric disorders) | 0 | 2
Unintended Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Venlafaxine Extended Release (ER) (N=269) | Venlafaxine Extended Release (ER) Plus Dialogues (N=268)
Asthenia (General disorders) | 14 | 19
Headache (General disorders) | 30 | 20
Infection (General disorders) | 17 | 12
Cardiovascular general (Cardiac disorders) | 28 | 27
Constipation (Gastrointestinal disorders) | 11 | 34
Diarrhea (Gastrointestinal disorders) | 8 | 15
Dry mouth (Gastrointestinal disorders) | 11 | 17
Nausea (Gastrointestinal disorders) | 27 | 42
Metabolic and nutritional general (Metabolism and nutrition disorders) | 9 | 15
Musculoskeletal general (Musculoskeletal and connective tissue disorders) | 9 | 15
Dizziness (Nervous system disorders) | 17 | 20
Insomnia (Nervous system disorders) | 36 | 38
Somnolence (Nervous system disorders) | 17 | 17
Respiratory general (Respiratory, thoracic and mediastinal disorders) | 45 | 43
Skin and appendages general (Skin and subcutaneous tissue disorders) | 23 | 27
Special senses general (Eye disorders) | 14 | 12
Urogenital general (Renal and urinary disorders) | 28 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.